CLINICAL TRIAL: NCT04323436
Title: A Double-blind, Placebo Controlled, Randomized, Phase II Study Evaluating the Efficacy and Safety of Capmatinib and Spartalizumab vs Capmatinib and Placebo as 1st Line Treatment for Advanced NSCLC Patients With MET exon14 Skipping Mutations
Brief Title: Study of Capmatinib and Spartalizumab/Placebo in Advanced NSCLC Patients With MET Exon 14 Skipping Mutations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study termination based on sponsor decision due to lack of tolerability observed with capmatinib and spartalizumab combination treatment when compared to data from capmatinib single agent studies
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CINC280J12201; 2019-003097-11 (EudraCT Number)
Record Dates: First submitted 2020-03-23; First posted 2020-03-26 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: capmatinib; spartalizumab; MET mutation; EGFR wild-type; ALK negative mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — spartalizumab; capmatinib

STUDY DESIGN:
Intervention Model Description: Run-in part: single arm, open-label.
  Randomized part: two-arms parallel assignment, double-blinded, placebo control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Run-in part (Experimental): capmatinib in combination with spartalizumab
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Randomized part - Arm 1 spartalizumab (Experimental): capmatinib in combination with spartalizumab
  Interventions: Drug: Spartalizumab; Drug: Capmatinib
- Randomized part - Arm 2 placebo (Experimental): capmatinib in combination with placebo
  Interventions: Drug: Capmatinib; Drug: spartalizumab placebo

INTERVENTIONS:
Drug: Spartalizumab — Concentrate for solution for infusion
  Other Names: PDR001
  Arms: Randomized part - Arm 1 spartalizumab; Run-in part
Drug: Capmatinib — Film-coated tablet
  Other Names: INC280
Drug: spartalizumab placebo — dextrose 5% in water (D5W) for infusion
  Other Names: PDR001 placebo
  Arms: Randomized part - Arm 2 placebo

SUMMARY:
A double-blind, placebo controlled, randomized, phase II study evaluating the efficacy and safety of capmatinib (INC280) and spartalizumab (PDR001) combination therapy versus capmatinib and placebo as first line treatment for locally advanced or metastatic non-small cell lung cancer (NSCLC) patients with MET exon 14 skipping (METΔex14) mutations

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of capmatinib in combination with spartalizumab in treatment naive patients with EGFR wild-type, ALK rearrangement negative advanced NSCLC, harboring METΔex14 mutations.

A run-in part (Part 1) was conducted to determine the anti-tumor activity and safety of capmatinib in combination with spartalizumab. Upon review of safety data and confirmation of anti-tumor activity in Part 1, the randomized part (Part 2) was planned to be initiated to compare the efficacy and safety of capmatinib plus spartalizumab to capmatinib plus placebo.

Combined treatment of METΔex14 mutated NSCLC with capmatinib and spartalizumab was expected to result in improved efficacy compared to each single agent due to direct targeting of an oncogenic driver (MET) as well as more efficient stimulation of an anti-tumor immune response than with PD-1 blockade alone.

The study enrollment was halted on 28-Jul-2021 per sponsor's decision. The enrollment halt decision was based on lack of tolerability observed in capmatinib and spartalizumab combination treatment in the run-in part (Part 1) of the trial.

Following the study enrollment halt during Part 1 (Run in Part), Part 2 was not initiated.

Immediately following the enrollment halt:

* All ongoing subjects were discontinued from spartalizumab treatment and continue to receive single agent capmatinib
* Enrolled subjects who had not started study treatment were to receive capmatinib single agent treatment from the start

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed locally advanced or metastatic NSCLC which is EGFR wild-type, ALK rearrangement negative and METΔex14 mutated
* No prior systemic therapy for advanced/metastatic disease (neo-adjuvant/adjuvant treatment completed > 12 months before relapse are permitted)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Measurable disease as per RECIST 1.1
* Known PD-L1 tumor expression status (applicable to Randomized part 2 only)

Key Exclusion Criteria:

* Prior treatment with a PD-1/PD-L1 inhibitor, MET inhibitor or HGF inhibitor
* Presence of symptomatic CNS metastases or requiring local CNS-directed therapy (radiotherapy or surgery), or increasing doses of corticosteroids 2 weeks prior to study entry
* Impaired cardiac function or clinically significant cardiac disease
* Presence or history of interstitial lung disease, non-infectious pneumonitis or interstitial pneumonitis, including clinically significant radiation pneumonitis
* History of allogenic bone marrow or solid organ transplant
* Radiotherapy to lung fields ≤ 4 weeks or to any other anatomic site ≤ 2 weeks prior to start of study treatment (palliative radiotherapy for bone lesions is allowed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Massachusetts General Hospital Liver and Kidney TX, Boston, Massachusetts, United States
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Montreal, Quebec, Canada
- France (3):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
- Germany (4):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Gerlingen
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Bologna, BO, Italy
- Novartis Investigative Site, Ōsaka-sayama, Osaka, Japan
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 15 investigative sites in 9 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed within 28 days prior to the first dose of study treatment. After screening, the treatment period started on Cycle 1 Day 1.
  The study enrollment was halted during the Run-in part per sponsor's decision. Following the study enrollment halt, spartalizumab treatment was discontinued and Part 2 was not initiated.
Groups:
- Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W: Capmatinib 400 mg orally twice daily (BID) in combination with spartalizumab 400 mg intravenously every 28 days (Q4W) in the run-in part.
- Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W: Capmatinib 400 mg orally twice daily (BID) in combination with spartalizumab 400 mg intravenously every 28 days (Q4W) in the randomized part.
- Randomized Part: Capmatinib 400 mg BID + Placebo: Capmatinib 400 mg orally twice daily (BID) in combination with spartalizumab matching placebo intravenously every 28 days (Q4W) in the randomized part.
Period: Overall Study
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Started | 31 | 0 | 0
Treated With Capmatinib + Spartalizumab | 28 | 0 | 0
Treated With Capmatinib Only (Immediately following the discontinuation of spartalizumab (and enrollment halt), enrolled subjects who had not started study treatment received capmatinib single agent treatment from the start.) | 3 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 31 | 0 | 0
Not completed — Adverse Event | 7 | 0 | 0
Not completed — Transfer to another clinical study or to other alternative treatment option | 8 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Progressive disease | 10 | 0 | 0
Not completed — Subject decision | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients to whom study treatment had been assigned and who received at least one dose of study treatment (i.e. at least one dose of any component of the study treatment that is capmatinib or spartalizumab). The randomized part of the study was not initiated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo | Total
Number analyzed (Participants) | 31 | 0 | 0 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (9.50) |  |  | 71.6 (9.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 0 | 0 | 16
  Male | 15 | 0 | 0 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23 | 0 | 0 | 23
  Black or African American | 1 | 0 | 0 | 1
  Asian | 6 | 0 | 0 | 6
  Unknown | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Run-in Part: Overall Response Rate (ORR) by Investigator Assessment as Per RECIST 1.1
Description: Tumor response was based on local investigator assessment as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 2 years and 4 months
Population: All patients to whom study treatment had been assigned and who received at least one dose of study treatment (i.e. at least one dose of any component of the study treatment that is capmatinib or spartalizumab) in the single arm run-in part. Patients were analyzed according to the treatment they were assigned to.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 31
percentage of participants | 35.5 [19.2 to 54.6]

2. Primary Outcome: Randomized Part: Progression-Free Survival (PFS) by BIRC as Per RECIST 1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. Tumor response based on blinded independent review committee (BIRC) assessment per RECIST v1.1.
Time Frame: Up to 6 years
Population: All patients to whom study treatment had been assigned and who received at least one dose of study treatment in the randomized part. The randomized part of the study was not initiated and data was not collected.
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Run-in Part: Number of Participants With Dose Reductions and Dose Interruptions of Capmatinib
Description: Number of participants with at least one dose reduction of capmatinib and number of participants with at least one dose interruption of capmatinib.
Time Frame: From first dose of capmatinib to last dose, up to 2.4 years
Population: All patients to whom study treatment had been assigned and who received at least one dose of capmatinib in the single arm run-in part. Patients were analyzed according to the treatment they were assigned to.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 31
Participants
  At least one dose reduction | 19
  At least one dose interruption | 20

4. Secondary Outcome: Run-in Part: Number of Participants With Dose Reductions and Dose Interruptions of Spartalizumab
Description: Number of participants with at least one dose reduction of spartalizumab and number of participants with at least one dose interruption of spartalizumab. Dose reductions were not allowed for spartalizumab.
Time Frame: From first dose of spartalizumab to last dose, up to 0.9 years
Population: All patients to whom study treatment had been assigned and who received at least one dose of spartalizumab in the single arm run-in part. Patients were analyzed according to the treatment they were assigned to.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 28
Participants
  At least one dose reduction | 0
  At least one dose interruption | 7

5. Secondary Outcome: Run-in Part: Dose Intensity of Capmatinib
Description: Dose intensity of capmatinib was calculated as actual cumulative dose in milligrams divided by duration of exposure in days.
Time Frame: From first dose of capmatinib to last dose, up to 2.4 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/day
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 31
mg/day | 595.9 (173.6)

6. Secondary Outcome: Run-in Part: Dose Intensity of Spartalizumab
Description: Dose intensity of spartalizumab was calculated as actual cumulative dose in milligrams divided by duration of exposure in days and then multiplied by the duration of one cycle (28 days).
Time Frame: From first dose of spartalizumab to last dose, up to 0.9 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/cycle
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 28
mg/cycle | 365.6 (51.5)

7. Secondary Outcome: Run-in Part: Disease Control Rate (DCR) by Investigator Assessment as Per RECIST 1.1
Description: DCR is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and non-CR/non-progressive disease (for subjects without target lesions). Tumor response was based on local investigator assessment per RECIST v1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression).
Time Frame: Up to approximately 2 years and 4 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 31
percentage of participants | 77.4 [58.9 to 90.4]

8. Secondary Outcome: Run-in Part: Progression-Free Survival (PFS) by Investigator Assessment as Per RECIST 1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on investigator assessment per RECIST v1.1. Progression is defined using RECIST v1.1 as at least 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: Up to approximately 2 years and 5 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 31
months | 16.5 [7.4 to NA] — Not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Run-in Part: Maximum Observed Plasma Concentration (Cmax) of Capmatinib
Description: Pharmacokinetic (PK) parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed plasma concentration following a dose.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: Patients in the capmatinib full pharmacokinetic analysis set (INC-FPAS) with an available value for the outcome measure. INC-FPAS consists of all patients who had an extensive PK sampling and provided a capmatinib evaluable PK profile on Cycle 3 Day 1.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 7
ng/mL | 2730 (74.3)

10. Secondary Outcome: Run-in Part: Time to Reach Maximum Plasma Concentration (Tmax) of Capmatinib
Description: PK parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) plasma concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 7
hours | 1.75 [1.00 to 3.92]

11. Secondary Outcome: Run-in Part: Area Under the Plasma Concentration-time Curve From Time Zero to the End of a Dosing Interval (AUCtau) of Capmatinib
Description: PK parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUCtau calculation. A dosing interval (tau) is defined as 12 hours. The portion of area under the curve between 8 hours and 12 hours post-dose was calculated by extrapolation based on terminal elimination slop.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 3
hr*ng/mL | 12900 (96.1)

12. Secondary Outcome: Run-in Part: Area Under the Plasma Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Capmatinib
Description: PK parameters were calculated based on capmatinib plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: pre-dose and 1, 2, 4 and 8 hours after morning dose on Cycle 3 Day 1. The duration of one cycle was 28 days.
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 7
hr*ng/mL | 10000 (61.8)

13. Secondary Outcome: Run-in Part: Maximum Observed Serum Concentration (Cmax) of Spartalizumab
Description: Pharmacokinetic (PK) parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-infusion and 1, 72, 168, 336 and 672 hours after completion of the spartalizumab infusion on Cycle 3 Day 1. The duration of the infusion was approximately 30 minutes. The duration of one cycle was 28 days.
Population: Patients in the spartalizumab full pharmacokinetic analysis set (PDR-FPAS) with an available value for the outcome measure. PDR-FPAS consists of all patients who had an extensive PK sampling and provided a spartalizumab evaluable PK profile on Cycle 3.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 9
µg/mL | 135 (28.4)

14. Secondary Outcome: Run-in Part: Time to Reach Maximum Serum Concentration (Tmax) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Median (Full Range); unit: hours
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 9
hours | 1.67 [0.917 to 164]

15. Secondary Outcome: Run-in Part: Area Under the Serum Concentration-time Curve From Time Zero to the End of a Dosing Interval (AUCtau) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUCtau calculation. A dosing interval (tau) is defined as 28 days.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 8
hr*µg/mL | 49700 (47.8)

16. Secondary Outcome: Run-in Part: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*µg/mL
Arm/Group | Run-in Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W
Number analyzed (Participants) | 9
hr*µg/mL | 52900 (64.6)

17. Secondary Outcome: Randomized Part: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause.
Time Frame: Up to 12 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Randomized Part: Number of Participants With Dose Reductions and Dose Interruptions of Capmatinib and Spartalizumab
Description: Number of participants with at least one dose reduction of capmatinib and spartalizumab and number of participants with at least one dose interruption of capmatinib and spartalizumab.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Randomized Part: Dose Intensity of Capmatinib and Spartalizumab
Description: Dose intensity is defined as the ratio of actual cumulative dose and duration of exposure.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Randomized Part: Progression-Free Survival (PFS) by Investigator Assessment as Per RECIST 1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. Tumor response based on investigator assessment per RECIST v1.1.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Randomized Part: Disease Control Rate (DCR) by BIRC and Investigator Assessment as Per RECIST 1.1
Description: DCR is defined as the percentage of participants with a best overall response of Complete Response (CR), Partial Response (PR), Stable Disease (SD), and non-CR/non-progressive disease (for subjects without target lesions). Tumor response based on BIRC and local investigator assessment per RECIST v1.1.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Randomized Part: Overall Response Rate (ORR) by BIRC and Investigator Assessment as Per RECIST 1.1
Description: ORR is defined as the percentage of participants with a best overall response of Complete Response (CR) and Partial Response (PR). Tumor response based on BIRC and local investigator assessment per RECIST v1.1.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Randomized Part: Duration of Response (DOR) by BIRC and Investigator Assessment as Per RECIST 1.1
Description: DOR is defined as the time from the date of first documented response (CR or PR) to the first documented progression per RECIST 1.1 or death due to any cause.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Randomized Part: Time to Response (TTR) by BIRC and Investigator Assessment as Per RECIST 1.1
Description: TTR is defined as the time from the date of start of treatment to the first documented response of either CR or PR, which must be subsequently confirmed, according to RECIST 1.1.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Randomized Part: Change From Baseline in EORTC QLQ-C30
Description: The European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) contains 30 items and is composed of both multi-item scales and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive, and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact) and a global health status/QoL scale. All scales and single-item measures range in score from 0 to 100. For the functional and the global QoL scales, a higher score indicates better health. For the symptom scales, a higher score indicates more symptom burden. The QLQ-C30 summary score (0-100) is calculated as the mean of 13 of the 15 QLQ-C30 scale and item scores (excluding global QoL and financial impact), with a higher score indicating a better health-related QoL.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Randomized Part: Change From Baseline in EORTC QLQ-LC13
Description: EORTC QLQ-LC13 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The five domains of the LC13 include pain, dyspnea, coughing and hemoptysis, and are based on their presence over the past week. All but the pain domain are scored on a 4 point Likert scale ranging from "not at all" to "very much". Pain score is based on its presence, hence yes or no. Scores are averaged and transformed to 0 to 100. A higher score indicates a higher presence of symptoms.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Randomized Part: Change From Baseline in EQ-5D-5L
Description: The EQ-5D-5L is a standardized measure of health utility that provides a single index value for one's health status. The EQ-5D-5L contains one item for each of five dimensions of health-related quality of life (HRQOL) (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Response options for each item vary from having no problems to extreme problems. Subject responses to the five dimensions of HRQOL reflect a specific health state that corresponds to a population preference weight for that state on a continuous scale of 0 (death) to 1 (perfect health). A visual analog scale (ranging from 0 to 100) is also included to capture subject's rating of their overall health status. Higher scores of the EQ-5D-5L represent better health states.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Randomized Part: Time to Definitive 10 Points Deterioration Symptom Scores for Pain in Chest, Coughing and Dyspnea Per QLQ-LC13 Questionnaire
Description: EORTC QLQ-LC13 is used in conjunction with the EORTC QLQ-C30 and provides information on an additional 13 items specifically related to lung cancer. The five domains of the LC13 include pain in chest, dyspnea, coughing and hemoptysis, and are based on their presence over the past week. All but the pain domain are scored on a 4 point Likert scale ranging from "not at all" to "very much". Pain score is based on its presence, hence yes or no. Scores are averaged and transformed to 0 to 100. A higher score indicates a higher presence of symptoms.
  The time to definitive 10 points deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10 points relative to baseline worsening of the corresponding scale score or death due to any cause.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

29. Secondary Outcome: Randomized Part: Time to Definitive Deterioration in Global Health Status/QoL, Shortness of Breath and Pain Per EORTC QLQ-C30
Description: The EORTC QLQ-C30 contains 30 items and is composed of both multi-item scales and single-item measures. These include 5 functional scales (physical, role, emotional, cognitive, and social functioning), 3 symptom scales (fatigue, nausea/vomiting, and pain), 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial impact) and a global health status/QoL scale. All scales and single-item measures range in score from 0 to 100. For the functional and the global QoL scales, a higher score indicates better health. For the symptom scales, a higher score indicates more symptom burden.
  The time to definitive 10 points deterioration is defined as the time from the date of randomization to the date of event, which is defined as at least 10 points relative to baseline worsening of the corresponding scale score or death due to any cause.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Randomized Part: Maximum Observed Concentration (Cmax) of Capmatinib and Spartalizumab
Description: Pharmacokinetic (PK) parameters calculated based on capmatinib and spartalizumab concentrations in plasma and serum, respectively, by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

31. Secondary Outcome: Randomized Part: Time to Reach Maximum Concentration (Tmax) of Capmatinib and Spartalizumab
Description: Pharmacokinetic (PK) parameters calculated based on capmatinib and spartalizumab concentrations in plasma and serum, respectively, by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) concentration following a dose.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

32. Secondary Outcome: Randomized Part: Area Under the Concentration-time Curve From Time Zero to the End of a Dosing Interval (AUCtau) of Capmatinib and Spartalizumab
Description: Pharmacokinetic (PK) parameters calculated based on capmatinib and spartalizumab concentrations in plasma and serum, respectively, by using non-compartmental methods.
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

33. Secondary Outcome: Randomized Part: Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Capmatinib and Spartalizumab
Description: as for outcome 32
Time Frame: Up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Randomized Part: Number of Participants With Anti-spartalizumab Antibodies
Description: Immunogenicity (IG) evaluated in serum samples. The assay to quantify and assess the IG was a validated homogeneous enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline (pre-dose), up to 6 years
Population: as for outcome 2
Arm/Group | Randomized Part: Capmatinib 400 mg BID + Spartalizumab 400 mg Q4W | Randomized Part: Capmatinib 400 mg BID + Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of spartalizumab+capmatinib (or capmatinib single agent for enrolled patients who had not started study treatment at the time of spartalizumab discontinuation) to 150 days after last dose of spartalizumab or 30 days after last dose of capmatinib, whichever was longer, up to approximately 2 years and 5 months.
Description: Patients were analyzed according to the treatment they actually received.
Groups:
- Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (Prior Discontinuing Spartalizumab): Capmatinib 400 mg BID in combination with spartalizumab 400 mg Q4W before the discontinuation of spartalizumab
- Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (After Discontinuing Spartalizumab): Capmatinib 400 mg BID in combination with spartalizumab 400 mg Q4W after the discontinuation of spartalizumab
- Run-in Part: Capmatinib 400mg BID Only: Immediately following the discontinuation of spartalizumab (and enrollment halt), enrolled subjects who had not started study treatment received capmatinib single agent treatment from the start
Arm/Group | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (Prior Discontinuing Spartalizumab) | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (After Discontinuing Spartalizumab) | Run-in Part: Capmatinib 400mg BID Only
All-Cause Mortality (participants affected / at risk) | 4/28 | 0/28 | 0/3
Serious Adverse Events (participants affected / at risk) | 11/28 | 8/28 | 1/3
Other Adverse Events (participants affected / at risk) | 25/28 | 18/28 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (Prior Discontinuing Spartalizumab) (N=28) | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (After Discontinuing Spartalizumab) (N=28) | Run-in Part: Capmatinib 400mg BID Only (N=3)
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
General physical health deterioration (General disorders) | 1 | 0 | 1
Medical device site haemorrhage (General disorders) | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0
Clostridium colitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Inferior vena cava syndrome (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (Prior Discontinuing Spartalizumab) (N=28) | Run-in Part: Capmatinib 400mg BID + Spartalizumab 400mg Q4W (After Discontinuing Spartalizumab) (N=28) | Run-in Part: Capmatinib 400mg BID Only (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 9 | 2 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 1
Chest pain (General disorders) | 2 | 1 | 1
Face oedema (General disorders) | 3 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 1
Oedema (General disorders) | 1 | 4 | 0
Oedema peripheral (General disorders) | 11 | 15 | 3
Pyrexia (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 8 | 6 | 1
Amylase increased (Investigations) | 3 | 4 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 6 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 1
Blood bilirubin increased (Investigations) | 2 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 4 | 0
Blood creatinine increased (Investigations) | 10 | 11 | 2
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 1
Lipase increased (Investigations) | 3 | 5 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Platelet count decreased (Investigations) | 2 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 1
Weight increased (Investigations) | 2 | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 1
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT04323436/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/36/NCT04323436/SAP_001.pdf